CLINICAL TRIAL: NCT00521521
Title: A Multicenter, Randomized, Phase II Study of the Combination of Docetaxel (TAXOTERE) and Concomitant Radiotherapy With or Without Cisplatin in Patients With Locally Advanced Head and Neck Cancer
Brief Title: Study of Combination Docetaxel and Radiotherapy With or Without Cisplatin to Treat Local Advanced Head and Neck Cancer
Acronym: TAX200006
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAX_FR1_236
Record Dates: First submitted 2007-08-27; First posted 2007-08-28 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Docetaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- docetaxel and cisplatin (Active Comparator)
  Interventions: Drug: docetaxel and cisplatin
- docetaxel (Experimental)
  Interventions: Drug: docetaxel

INTERVENTIONS:
Drug: docetaxel and cisplatin
  Arms: docetaxel and cisplatin
Drug: docetaxel
  Arms: docetaxel

SUMMARY:
To evaluate the efficacy of the concomitant combination of radiotherapy and docetaxel with or without cisplatin in terms of objective response rates (WHO criteria).

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced head and neck cancer (T3 and T4 tumors), epidermoid, histologically proven without metastasis; the primitive site of which is the oral cavity, the oropharynx, the hypopharynx or the larynx.
* Locally advanced tumors which are inoperable, or operable but the patient refuses surgery.
* Age ≥ 18 years and ≤ 70 years.
* PS < 2.
* Satisfactory hematological, hepatic and renal functions: (PN ≥ 2000/mm3, platelet count ≥ 100,000/mm3, hemoglobin ≥ 10g/dl, serum creatinine ≤ 120 µmol/l or creatinine clearance ≥ 60 ml/mn, normal total bilirubin, AST (SGOT) and ALT (SGPT) ≤ 2.5 x the upper limit of normal (ULN) of each center, PAL ≤ 5 x LNS; patients with AST or ALT > 1.5 x LNS combined with PAL > 2.5 x LNS will not be eligible for this trial.

Exclusion Criteria:

* Any metastases (other than cervical ganglia).
* Cancer of the cavum and the facial structure.
* Any previous chemotherapy or radiotherapy, irrespective of the reason.
* Any surgery for epidermoid carcinoma in the upper aerodigestive tracts.
* Weight loss ≥10% of total body weight during the last 3 months.
* Any other previous cancer excepting in situ or cutaneous cervical cancer (spinocellular or basocellular).
* Pregnant or nursing women; women of childbearing potential must use an appropriate method of contraception.
* Poorly controlled progressive infection.
* Peripheral neuropathy with NCI grade ≥ 2.
* Neurological or psychiatric disease (dementia, seizures, etc.) that is not compatible with good understanding and sufficient compliance with treatment.
* Any other poorly controlled progressive disease, such as heart failure, symptomatic cardiac rhythm disorders, progressive angina pectoris, or respiratory impairment.
* Any other concomitant investigational treatment.
* Any other concomitant anticancer treatment.
* Allergy to polysorbate 80.
* Definitive formal contraindication to corticosteroids.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2001-07; Primary Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Objective response rates | evaluated 8 weeks after the end of radiotherapy

SECONDARY OUTCOMES:
Duration of the responses and overall survival | time until progression

CONTACTS AND LOCATIONS:
Overall Officials: Marie SEBILLE, Dr., Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Paris, France